CLINICAL TRIAL: NCT02839941
Title: An Open-label Study to Evaluate the Effect of Iguratimod Concomitant With Conventional Immunosuppressive Drugs on Preventing Antibody-induced Rejection in Human Leukocyte Antigen(HLA) Highly Mismatched Kidney Transplant Recipients
Brief Title: Iguratimod in Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT-2016-1
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — iguratimod; Mycophenolic Acid; Tacrolimus; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experiment (Experimental)
  Interventions: Drug: Iguratimod; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Glucocorticoids
- Control (Sham Comparator)
  Interventions: Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Glucocorticoids

INTERVENTIONS:
Drug: Iguratimod — Subjects will receive iguratimod orally, twice a day, for consecutive 52 weeks
  Arms: experiment
Drug: Mycophenolate mofetil — All subjects will receive mycophenolate mofetil for consecutive 52 weeks
Drug: Tacrolimus — All subjects will receive tacrolimus for consecutive 52 weeks
Drug: Glucocorticoids — All subjects will receive glucocorticoids for consecutive 52 weeks

SUMMARY:
The objective of the study is to evaluate the effect of iguratimod concomitant with conventional immunosuppressive drugs on preventing antibody-induced rejection in HLA Highly mismatched Kidney Transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥18, <65 years
* At least 2 weeks post kidney transplantation from deceased or living donor
* Stable renal graft function, i.e., serum creatinine undulation for 3 consecutive test <±10%
* Serum creatinine<1.5×upper limits of normal(ULN)
* Number of HLA mismatches ≥ 4
* Panel Reactive Antibody(PRA) value pre-transplantation <10%
* Concentration of conventional immunosuppressive drugs reach target ranges
* Subjects are willing to participate in the study, fully informed, and sign informed consent form(ICF)
* Women of childbearing potential (WOCBP) must have a negative pregnancy test within 24 hours prior to the start of study medication, and agree to use an acceptable method to avoid pregnancy for the entire study period and for up to 3 months after the last dose of study medication.

Exclusion Criteria:

* Pregnant or nursing women
* Currently clinical acute rejection;
* Graft function hasn't recovered for delayed graft function (DGF), or primary non-function (PNF)
* Second or subsequent kidney transplant or multi-organ recipients (e.g. kidney and pancreas)
* Subjects with Liver failure
* Abnormal hepatic, renal and hematopoietic function,

  1. Alanine transaminase(ALT), Aspartate transaminase(AST)>1.5×ULN
  2. White blood cell(WBC)<3.5×10^9/L
  3. Hemoglobin(HGB)<80 g/L
  4. Platelet count(PLT)<80×10^9/L.
* Severe clinically relevant disease,

  1. Abnormality in chest X ray image, such as Tuberculosis, Pulmonary interstitial fibrosis, or symptom or physical sign of clinical significance
  2. Serious cardiovascular, hepatic, hematological, endocrinal disease, or malignancy 3）History of serious cardiovascular, hepatic, hematological, endocrinal disease, or malignancy

  4) Immunodeficiency, uncontrolled active infection, and active gastrointestinal disease.
* Women or men of childbearing potential plan to be pregnant recently;
* Allergic with study drug, or excipient
* Subject with psychiatric illness, which may put him/her into unacceptable risk in the opinion of investigators
* Has received or is receiving Rituximab treatment
* Iguratimod treatment within 1 week pre-transplantation, or during screening period
* Received live vaccines in the previous 3 months, or plan to receive live vaccines during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Biopsy-proven acute rejection rates | 0-52 week
Survival of transplanted kidney | 52 week

SECONDARY OUTCOMES:
Donor Specific Antibody(DSA) level compared to baseline | 52 week
Graft renal function | 52 week
Adverse event | 0-52 week

CONTACTS AND LOCATIONS:
Overall Officials: Min Gu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No